CLINICAL TRIAL: NCT01546571
Title: A Multicenter, Double-blind, Placebo-controlled, Adaptive Phase 3 Trial of POL-103A Polyvalent Melanoma Vaccine in Post-resection Melanoma Patients With a High Risk of Recurrence
Brief Title: Study of a Melanoma Vaccine in Stage IIb, IIc, and III Melanoma Patients
Acronym: MAVIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After interim analysis the study was halted to redesign a pivotal trial.
Sponsor: Polynoma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 103A-301
Record Dates: First submitted 2012-02-26; First posted 2012-03-07 (Estimated); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- POL-103A without API (Placebo Comparator)
  Interventions: Biological: POL-103A without API
- POL-103A (Experimental)
  Interventions: Biological: POL-103A

INTERVENTIONS:
Biological: POL-103A — POL-103A is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs
  Arms: POL-103A
Biological: POL-103A without API — Placebo is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs
  Arms: POL-103A without API

SUMMARY:
The purpose of this study is to determine how safe and how well POL-103A works in preventing the relapse of melanoma after patients who have undergone surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage IIb, IIc, III melanoma
* Surgical resection within 90 days of first dosing
* Persons with positive sentinel nodes must have a complete lymphadenectomy
* ECOG performance status 0 or 1

Exclusion Criteria:

* Any prior melanoma treatment other than surgery or regional irradiation
* Use of biologic response modifiers within 60 days of first dosing
* Subjects with history of other malignancy within past 5 years (with exceptions)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Slingluff, M.D., Principal Investigator — University of Virginia Hospital
Locations (65):
- United States (59):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - City of Hope National Medical Center, Duarte, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Sutter Cancer Center, Sacramento, California
  - St. Mary's Hospital & Medical Center Department of Pathology, San Francisco, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - The Melanoma Center at the Washington Cancer Institute, Washington D.C., District of Columbia
  - GenesisCare USA of Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center-Orlando, Orlando, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Advocate Medical Group, Niles, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Central Kentucky Research Associates, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Harry & Jeanette Weinberg Cancer Institute @ Franklin Square, Baltimore, Maryland
  - Ascension Providence Hospital, Southfield, Michigan
  - University of Minnesota Masonic Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Mayo Clinic Rochester, Rochester, Minnesota
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center / Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center/ Hackensack Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University School of Medicine, Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Premier Health Partners Clinical Trials Research Alliance, Dayton, Ohio
  - Independence Family Health Center (Cleveland Clinic), Independence, Ohio
  - Hillcrest Hospital (Cleveland Clinic), Mayfield Heights, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson Medical Oncology, Philadelphia, Pennsylvania
  - McGlinn Cancer Institute, Reading Hospital, West Reading, Pennsylvania
  - The West Clinic P.C. d/b/a West Cancer Center, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Cancer Solutions, Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - The Huntsman Cancer Institute, University of Utah Health Care, Salt Lake City, Utah
  - University of Virginia Hospital, Charlottesville, Virginia
  - Inova Schar Cancer Center, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Multicare Institute for Research & Innovation, Tacoma, Washington
- Canada (6):
  - BCCA Vancouver Island Cancer Centre, Victoria, British Columbia
  - Durham Regional Cancer Centre, Oshawa, Ontario
  - Princess Margaret Hospital, Department of Medical Oncology, Toronto, Ontario
  - CISSS de la Montérégie - Centre, Greenfield Park, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec, Québec

REFERENCES:
- [Derived] Slingluff CL, Lewis KD, Andtbacka R, Hyngstrom J, Milhem M, Markovic SN, Bowles T, Hamid O, Hernandez-Aya L, Claveau J, Jang S, Philips P, Holtan SG, Shaheen MF, Curti B, Schmidt W, Butler MO, Paramo J, Lutzky J, Padmanabhan A, Thomas S, Milton D, Pecora A, Sato T, Hsueh E, Badarinath S, Keech J, Kalmadi S, Kumar P, Weber R, Levine E, Berger A, Bar A, Beck JT, Travers JB, Mihalcioiu C, Gastman B, Beitsch P, Rapisuwon S, Glaspy J, McCarron EC, Gupta V, Behl D, Blumenstein B, Peterkin JJ. Multicenter, double-blind, placebo-controlled trial of seviprotimut-L polyvalent melanoma vaccine in patients with post-resection melanoma at high risk of recurrence. J Immunother Cancer. 2021 Oct;9(10):e003272. doi: 10.1136/jitc-2021-003272. PMID 34599031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A (dose finding) was competitive enrollment from 6/1/2012 to 10/16/2013. Part B1 of the protocol was competitive enrollment from 1/1/2015 to 8/16/2016. The study was halted prior to Part B2. Types of sites range from clinical oncologist, dermatological and surgical oncologist.
Groups:
- Part A POL-103A 40 Micrograms/Dose; Part A POL-103A 100 Micrograms/Dose: POL-103A: Placebo is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
- Part A Without API; Part B1 POL-103A Without API: POL-103A without API: Placebo is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
- Part B1 POL-103A 40 Micrograms/Dose: POL-103A: POL-103A is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
Period: Overall Study
Arm/Group | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A 100 Micrograms/Dose | Part A Without API | Part B1 POL-103A 40 Micrograms/Dose | Part B1 POL-103A Without API
Started | 52 | 52 | 53 | 230 | 117
Completed | 29 | 29 | 7 | 141 | 74
Not Completed | 23 | 23 | 46 | 89 | 43
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0
Not completed — assigned placebo in Part A | 0 | 0 | 22 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 20 | 18 | 15 | 73 | 37
Not completed — Withdrawal by Subject | 1 | 2 | 4 | 9 | 2
Not completed — Intercurrent Illness | 1 | 2 | 0 | 0 | 0
Not completed — Other Cancers | 0 | 0 | 0 | 3 | 1
Not completed — Other | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A POL-103A 40microgram/Dose; Part A POL-103A 100 Microgram/Dose; Part A POL-103A Without API; Part B1 POL-103A Without API: POL-103A without API: Placebo is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
- Part B1 POL-103A: POL-103A: POL-103A is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
- Total: Total of all reporting groups
Arm/Group | Part A POL-103A 40microgram/Dose | Part A POL-103A 100 Microgram/Dose | Part A POL-103A Without API | Part B1 POL-103A | Part B1 POL-103A Without API | Total
Number analyzed (Participants) | 52 | 52 | 53 | 230 | 117 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (9.74) | 53.8 (12.73) | 55.8 (14.90) | 56.3 (12.73) | 55.8 (13.73) | 56.1 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 20 | 96 | 52 | 202
  Male | 36 | 34 | 33 | 134 | 65 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 7 | 4 | 16
  Not Hispanic or Latino | 50 | 50 | 52 | 222 | 113 | 487
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  North America | 52 | 52 | 53 | 230 | 117 | 504

OUTCOME MEASURES:

1. Primary Outcome: Part B1: Recurrence Free Survival (RFS)
Description: This is an event driven trial. Recurrence-free survival time (RFS) is computed from the earliest of the date of recurrence or death or, if without recurrence or death, the date last assessed for recurrence without diagnosis of recurrence (censored). The date of recurrence is specified as the first date a recurrence is suspected, which is later confirmed by biopsy.
Time Frame: 432 events or 8 years and 10 months
Population: Overall Status of patients at the end of the study. This is applicable to Part B1 only. Study was halted prior to Part B2.
Measure: Count of Participants; unit: Participants
Groups:
- Part B1 POL-103A-Stage IIB/IIC; Part B1 POL-103A-IIIA; Part B1 POL-103A -IIIB/IIIC; Part B1 POL-103A All Randomized: POL-103A: POL-103A is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs
- Part B1 POL-103A Without API-IIB/IIC; Part B1 POL-103A Without API-IIIA; Part B1 POL-103A Without API-IIIB/IIIC; Part B1 POL-103A Without API-All Randomized: POL-103A without API: Placebo is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs
Arm/Group | Part B1 POL-103A-Stage IIB/IIC | Part B1 POL-103A Without API-IIB/IIC | Part B1 POL-103A-IIIA | Part B1 POL-103A Without API-IIIA | Part B1 POL-103A -IIIB/IIIC | Part B1 POL-103A Without API-IIIB/IIIC | Part B1 POL-103A All Randomized | Part B1 POL-103A Without API-All Randomized
Number analyzed (Participants) | 74 | 37 | 69 | 34 | 87 | 46 | 230 | 117
Participants
  Participants with recurrence | 32 | 20 | 18 | 13 | 51 | 23 | 101 | 56
  Participants censored | 42 | 17 | 51 | 21 | 36 | 23 | 129 | 61

2. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight MW) Range 1 [0,20)
Description: For Part A, immunogenicity of the vaccine was based on anti-melanoma IgG/IgM antibody response at week 10 compared to week 0. A positive result by Western Blot was considered an immunogenic response to study treatment. The response for each participant was calculated based on the average percent change in intensity across these Bins. The definition of response in each participant was the average percent change: > 0% (meaning any change), or > 5, 10, 15, 20, and 25%. The bands having data in each Bin is the unit of analysis in each Bin and in all cases corresponds to the number of participants having bands in that Bin. No participant had multiple bands in a single Bin.
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for WM range 1.
Population: The definition of response in each participant was the average percent change: > 0% (meaning any change), or > 5, 10, 15, 20, and 25%.
  The bands having data in each Bin is the unit of analysis in each Bin and in all cases corresponds to the number of participants having bands in that Bin.
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Groups:
- Part A POL-103A 100 Micrograms/Dose; Part A POL-103A 40 Micrograms/Dose; Part A POL-103A Without API: POL-103A without API: Placebo is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 20 | 17 | 27
percentage of change in bands | 6.8 (44.9) | 7.3 (26.1) | -1.8 (29.8)

3. Secondary Outcome: Part B1: Overall Survival (OS)
Description: Overall survival (OS) analyses were based on the ITT analysis set; OS was defined as the duration from randomization until death. If the patient was alive, OS was censored at the earliest date the participant was known to be alive or the date of data cutoff.
Time Frame: Overall survival (OS) was measured from randomization until death from any cause, assessed up to 76 months.
Population: Part B1 participants randomized to seviprotimut-L 40 μg or placebo. Part B2 was not initiated.
Measure: Count of Participants; unit: Participants
Groups:
- POL-103A Without API: POL-103A without API: Placebo is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
- POL-103A: POL-103A: POL-103A is administered intradermally, divided into 4 injections (0.2 mL each injection) into the volar surface of forearms and into the anterior upper thighs. A total of 15 dosing visits over 2 years.
Arm/Group | POL-103A Without API | POL-103A
Number analyzed (Participants) | 117 | 230
Participants | 97 | 201
Statistical Analysis 1: Comparison: POL-103A Without API vs POL-103A; Test type: Other; Hazard Ratio (HR) = .44

4. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 2 [20,28)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 20 | 29 | 28
percentage of change in bands | 0.4 (22.3) | 12.0 (38.4) | -6.2 (16.3)

5. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 3 [28,36)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 19 | 21 | 24
percentage of change in bands | 14.8 (74.2) | 9.3 (32.9) | 0.5 (35.1)

6. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 4 [36,44)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 27 | 21 | 28
percentage of change in bands | 5.3 (24.6) | 7.6 (20.7) | 8.5 (43.5)

7. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 5 [44,53)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 27 | 27 | 36
percentage of change in bands | 1.3 (23.1) | 9.5 (43.3) | 10.3 (33.0)

8. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 6 [53,62)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 74 | 10 | 10
percentage of change in bands | -12.7 (19.5) | 18.8 (49.0) | 14.4 (29.1)

9. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 7 [62,72)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 21 | 20 | 21
percentage of change in bands | 6.8 (24.4) | 5.5 (22.7) | 7.9 (28.4)

10. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 8 [72,83)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 31 | 33 | 32
percentage of change in bands | -0.0 (18.2) | 0.4 (16.8) | 10.5 (35.9)

11. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 9 [83,94)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 16 | 17 | 18
percentage of change in bands | -0.8 (24.3) | 16.8 (25.6) | 5.9 (34.7)

12. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 10 [94,105)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 24 | 22 | 30
percentage of change in bands | 13.7 (31.4) | 4.0 (21.4) | 9.9 (27.5)

13. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 11 [105,118)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 11
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 28 | 23 | 25
percentage of change in bands | 5.1 (23.8) | 1.0 (19.3) | 5.0 (31.7)

14. Primary Outcome: Part A:To Evaluate the Biological Activity of Seviprotimut-L in Patients With Molecular Weight (MW) Range 12 [118,Inf)
Description: as for outcome 2
Time Frame: Serum was collected for Western blot testing and analysis on Day 0 (baseline) and at Week 10 for MW range 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change in bands
Arm/Group | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A Without API
Number analyzed (Participants) | 12 | 7 | 9
percentage of change in bands | 2.3 (15.9) | -5.3 (20.1) | -15.5 (26.9)

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from study treatment administration to 30 days following the last dose of study treatment-up to 24 months. All-Cause Mortality was assessed from treatment administration up to 8 years and 10 months.
Description: TEAE: AE b/w treatment (Tx) and 30 days post last dose, 2) AE started prior to Tx but worsened after Tx, 3) AE with partial onset/stop dated after 1st Tx and partial onset date did not definitely place AE before start date of Tx, 4) AE with missing onset date. AEs graded according to NCI Common Terminology Criteria for AEs. Participant counted once in most severe category w/multiple TEAEs reported; and once in closest related category when multiple TEAEs reported.
Arm/Group | Part A POL-103A 40 Micrograms/Dose | Part A POL-103A 100 Micrograms/Dose | Part A POL-103A Without API | Part B1 POL-103A | Part B1 POL-103A Without API
All-Cause Mortality (participants affected / at risk) | 12/52 | 12/52 | 6/53 | 29/230 | 20/117
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/53 | 0/230 | 0/117
Other Adverse Events (participants affected / at risk) | 48/52 | 51/52 | 51/53 | 212/230 | 113/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A POL-103A 40 Micrograms/Dose (N=52) | Part A POL-103A 100 Micrograms/Dose (N=52) | Part A POL-103A Without API (N=53) | Part B1 POL-103A (N=230) | Part B1 POL-103A Without API (N=117)
Injection site erythema (Infections and infestations) | 13 (87) | 16 (267) | 18 (261) | 73 (583) | 50 (307)
Fatigue (General disorders) | 17 (24) | 13 (19) | 16 (19) | 64 (97) | 42 (64)
Injection site pruritus (Infections and infestations) | 4 (10) | 8 (54) | 4 (17) | 46 (374) | 16 (64)
Headache (Nervous system disorders) | 7 (8) | 7 (8) | 4 (6) | 34 (56) | 23 (33)
Injection site pain (Infections and infestations) | 1 (2) | 4 (24) | 3 (10) | 32 (319) | 13 (153)
Nausea (General disorders) | 8 (13) | 5 (8) | 5 (5) | 31 (40) | 11 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (17) | 5 (5) | 3 (3) | 21 (26) | 18 (21)
Diarrhea (Gastrointestinal disorders) | 7 (10) | 6 (7) | 2 (2) | 20 (26) | 13 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2) | 3 (3) | 13 (14) | 13 (14)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (7) | 6 (7) | 2 (3) | 16 (21) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (6) | 1 (1) | 19 (22) | 15 (20)
Cataract (Eye disorders) | 4 (5) | 3 (5) | 1 (1) | 7 (7) | 9 (9)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1) | 8 (10) | 7 (8)
Injection site urticaria (General disorders) | 6 (108) | 8 (116) | 5 (51) | 5 (52) | 0 (0)
Injection site nodule (General disorders) | 1 (1) | 5 (20) | 6 (39) | 5 (8) | 2 (5)
Influenza like illness (General disorders) | 4 (8) | 2 (2) | 8 (12) | 13 (26) | 8 (9)
Oedema Peripheral (General disorders) | 4 (5) | 3 (3) | 1 (1) | 17 (21) | 5 (5)
Injection site swelling (General disorders) | 2 (4) | 3 (24) | 3 (13) | 15 (97) | 6 (19)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (18) | 6 (8)
Injection site induration (General disorders) | 3 (43) | 3 (38) | 2 (32) | 9 (28) | 3 (66)
Peripheral swelling (General disorders) | 5 (7) | 1 (1) | 1 (1) | 3 (3) | 4 (5)
Injection site rash (General disorders) | 3 (4) | 1 (18) | 2 (6) | 8 (15) | 4 (7)
Pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 5 (8) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6) | 1 (1) | 26 (27) | 9 (13)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2) | 3 (4) | 13 (15) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (4) | 15 (15) | 14 (18)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 4 (4) | 13 (15) | 10 (12)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 7 (10) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (3) | 3 (5) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 7 (7) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 4 (5) | 16 (22) | 11 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 1 (1) | 13 (16) | 8 (8)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 5 (6) | 2 (2) | 16 (21) | 6 (9)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 2 (2) | 5 (7) | 15 (22) | 4 (4)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (7) | 3 (4) | 1 (1) | 9 (10) | 3 (4)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 2 (4) | 9 (11) | 3 (6)
Dizziness (Nervous system disorders) | 5 (5) | 7 (7) | 1 (1) | 13 (14) | 7 (8)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 9 (9) | 7 (10)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (7)
Insomia (Psychiatric disorders) | 4 (7) | 5 (7) | 3 (3) | 12 (16) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 10 (11) | 7 (8)
Haematuria (Renal and urinary disorders) | 5 (6) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 0 (0) | 8 (8) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 9 (10) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8) | 5 (6) | 4 (4) | 22 (27) | 8 (9)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 3 (4) | 26 (26) | 4 (7) | 15 (37) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 6 (9)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7) | 2 (2) | 8 (9) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 8 (9) | 3 (3)
Lymphoedema (Vascular disorders) | 3 (3) | 2 (3) | 4 (4) | 9 (10) | 6 (8)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 15 (17) | 4 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 (7) | 1 (1) | 3 (3) | 6 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT01546571/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT01546571/SAP_001.pdf